CLINICAL TRIAL: NCT03234712
Title: A Phase 1 Study Evaluating the Safety, Pharmacokinetics, and Anti-tumor Activity of ABBV-321 in Subjects With Advanced Solid Tumors Associated With Overexpression of the Epidermal Growth Factor Receptor (EGFR)
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Anti-tumor Activity of ABBV-321 in Subjects With Advanced Solid Tumors Associated With Overexpression of the Epidermal Growth Factor Receptor (EGFR)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-438
Record Dates: First submitted 2017-07-27; First posted 2017-07-31 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Advanced Solid Tumors Cancer
Keywords: Advanced Solid Tumors; Epidermal Growth Factor Receptor (EGFR); Squamous cell carcinoma of the head and neck (HNSCC); non-small cell lung cancer (NSCLC); Glioblastoma (GBM); Cancer; overexpression of Epidermal Growth Factor Receptor (EGFR)
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma, Non-Small-Cell Lung; Glioblastoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABBV-321 (Experimental): ABBV-321 will be administered via intravenous infusion at escalating dose levels until the maximum tolerated dose is reached and a recommended Phase 2 dose is determined.
  Interventions: Drug: ABBV-321

INTERVENTIONS:
Drug: ABBV-321 — Intravenous infusion
  Other Names: Serclutamab Talirine

SUMMARY:
This is an open-label, Phase 1, dose-escalation study to determine the maximum tolerated dose (MTD) and the recommended phase two dose (RPTD), and to assess the safety, preliminary efficacy, and pharmacokinetic (PK) profile of ABBV-321 for participants with advanced solid tumors likely to overexpress the epidermal growth factor receptor (EGFR). The study will consist of 2 phases: Dose Escalation Phase and Expansion Phase.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Histologically or cytologically confirmed solid tumor of one of the following types associated with overexpression of Epidermal Growth Factor Receptor (EGFR). (For Expansion Phase: Subjects must have EGFR overexpression demonstrated by central assessment or Sponsor selected test).

Dose Escalation Phase:

* Colorectal cancer (CRC), Glioblastoma (GBM), squamous cell carcinoma of the head and neck (HNSCC), non-small cell lung cancer (NSCLC), bladder, cervical, esophageal, kidney or sarcoma.
* Participants must have disease that has progressed on prior treatment and is not amenable to surgical resection or other approved therapeutic options with curative intent. Participants must not be eligible for, or has refused further therapy that is likely to provide a survival benefit.
* Must have measureable disease as per RECIST Version 1.1 or RANO (for GBM).
* Minimum life expectancy of at least 12 weeks.

Expansion Phase (Solid Tumor Cohort):

* Histologically or cytologically confirmed advanced solid tumor.
* Participants must have disease that has progressed on prior treatment and is not amenable to surgical resection or other approved therapeutic options with curative intent.
* Must have measureable disease as per RECIST Version 1.1.
* Minimum life expectancy of at least 12 weeks.

Expansion Phase (GBM Cohort Only):

* Participant has recurrent primary (de novo) glioblastoma histologically confirmed at any time from initial diagnosis through latest recurrence.
* Participant has recurrent GBM per Response Evaluation in Neuro-Oncology (RANO) requirements.
* Tumor is measurable according to RANO criteria.

Exclusion Criteria:

* Active uncontrolled infection National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE Grade greater than or equal to 3).
* New York Heart Association (NYHA) Class III or IV heart failure and/or ejection fraction of < 40% as measured by echocardiogram at screening.
* Unstable angina pectoris or cardiac ventricular arrhythmia.
* Myocardial infarction or cerebrovascular accident (CVA) within 6 months.
* Documented history of capillary leak syndrome within 6 months of study enrollment.
* Grade 2 or higher peripheral edema, ascites, pleural, or pericardial effusion within 4 weeks of study enrollment or any history of recurrent grade 2 or higher effusions requiring ongoing drainage.
* Active keratitis or current corneal disorder.
* Laser-assisted in situ keratomileusis (LASIK) procedure within the last 1 year or cataract surgery within the last 3 months.
* Major surgery (including opening of the abdomen, chest) within 21 days of the first dose of study drug.
* Uncontrolled metastases from an extracranial solid tumor to the central nervous system (CNS). Participants with brain metastases from an extracranial solid tumor are eligible after definitive therapy provided they are asymptomatic for at least 2 weeks prior to first dose of ABBV-321.
* No history of medical condition resulting in nephrotic range proteinuria.
* Participants must not have been treated in anticancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal therapy, biologic therapy or investigational anti-cancer therapy within a period of 21 days or herbal anticancer therapy within 7 days prior to the first dose of study drug.
* For approved targeted small molecules, a washout period of 5 half-lives is adequate (no washout period required for subjects currently on erlotinib)
* Participant must not have been in more than three lines of systemic cytotoxic therapy (excluding adjuvant and neoadjuvant therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
AUCt for ABBV-321 | Up to 78 days post dose
  Area Under the Plasma Concentration-time Curve from Time 0 to the Time of the Last Measurable Concentration (AUCt) for ABBV-321
AUC∞ for ABBV-321 | Up to 78 days post dose
  AUC∞ is the area under the plasma concentration-time curve from Time 0 to infinite time.
Tmax of ABBV-321 | Up to 78 days post dose
  Time to Cmax (Tmax) of ABBV-321
Terminal phase elimination rate constant (β) for ABBV-321 | Up to 78 days post dose
  Terminal phase elimination rate constant (β)
Cmax of ABBV-321 | Up to 78 days post dose
  Maximum observed plasma concentration (Cmax) of ABBV-321
Dose Escalation Phase: Recommended Phase 2 dose (RPTD) for ABBV-321 | Minimum first cycle of dosing (up to 28 days)
  The RPTD will be determined using available safety and pharmacokinetics data upon completion of the Dose Escalation Phase
t1/2 for ABBV-321 | Up to 78 days post dose
  Terminal elimination half-life (t1/2)
Dose Escalation Phase: Maximum tolerated dose (MTD) of ABBV-321 | Minimum first cycle of dosing (up to 28 days)
  The MTD of ABBV-321 will be determined during the dose escalation phase of the study.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to approximately 5 years
  PFS is defined as the number of days from the first dose date to the earliest date of disease progression per RECIST 1.1 or RANO criteria or death, whichever occurred first.
Duration of Response (DOR) | Up to approximately 5 years
  DOR for a given participant is defined as the number of days from the day CR or PR (whichever is recorded first) occurred to the earliest date of disease progression per RECIST 1.1 or RANO criteria or death, whichever occurred first.
Disease Control Rate (DCR) | Up to 5 years
  DCR is defined as the proportion of participants with objective evidence of complete response (CR), partial response (PR) or stable disease (SD); a participants best overall response assignment of SD must be maintained for at least 6 weeks since the first dose date of study drug.
Time to progression (TTP) | Up to approximately 5 years
  TTP is defined as the number of days from the first dose date to the earliest date of disease progression per RECIST version 1.1 or RANO criteria.
Change from Baseline in QTcF | Up to 61 days post dose
  QT interval measurement corrected by Fridericia's formula (QTcF) change from baseline
Overall Survival (OS) | Up to approximately 5 years
  OS is defined as number of days from the date of the first dose to the date of death for all dosed participants. For participants who are not deceased, the data will be censored at the last known date to be alive.
Objective response rate (ORR) | Up to 5 years
  ORR is defined as the proportion of participants with a response of partial response (PR) or better; Response Assessment in Neuro-Oncology (RANO) criteria will be used for glioblastoma (GBM) participants, and Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria will be used for all other participants.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (18):
- United States (14):
  - Highlands Oncology Group /ID# 166132, Springdale, Arkansas
  - The Angeles Clinic and Researc /ID# 166133, Los Angeles, California
  - University of California, Davis Comprehensive Cancer Center /ID# 215012, Sacramento, California
  - Northwestern University Feinberg School of Medicine /ID# 165191, Chicago, Illinois
  - University of Chicago /ID# 166064, Chicago, Illinois
  - Northshore University Health System Dermatology Clinical Trials Unit /ID# 201095, Skokie, Illinois
  - University of Kentucky Markey Cancer Center /ID# 217665, Lexington, Kentucky
  - Dana-Farber Cancer Institute /ID# 212920, Boston, Massachusetts
  - Washington University-School of Medicine /ID# 214955, St Louis, Missouri
  - Columbia Univ Medical Center /ID# 167184, New York, New York
  - Stony Brook University Hospital /ID# 216976, Stony Brook, New York
  - Duke University Medical Center /ID# 166135, Durham, North Carolina
  - Lifespan Cancer Institute at Rhode Island Hospital /ID# 168600, Providence, Rhode Island
  - South Texas Accelerated Research Therapeutics /ID# 166134, San Antonio, Texas
- Australia (3):
  - Northern Cancer Institute /ID# 166138, St Leonards, New South Wales
  - Monash Health /ID# 217435, Clayton, Victoria
  - Austin Hospital /ID# 166137, Heidelberg, Victoria
- Sheba Medical Center /ID# 166398, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carneiro BA, Papadopoulos KP, Strickler JH, Lassman AB, Waqar SN, Chae YK, Patel JD, Shacham-Shmueli E, Kelly K, Khasraw M, Bestvina CM, Merrell R, Huang K, Atluri H, Ansell P, Li R, Jin J, Anderson MG, Reilly EB, Morrison-Thiele G, Patel K, Robinson RR, Aristide MRN, Gan HK. Phase I study of anti-epidermal growth factor receptor antibody-drug conjugate serclutamab talirine: Safety, pharmacokinetics, and antitumor activity in advanced glioblastoma. Neurooncol Adv. 2022 Dec 21;5(1):vdac183. doi: 10.1093/noajnl/vdac183. eCollection 2023 Jan-Dec. PMID 36814898